CLINICAL TRIAL: NCT03265470
Title: The Potential Renal Protective Effect of Intravenous Dexmedetomidine for Patients During Radical Cystectomy
Brief Title: Renal Protection of Intravenous Dexmedetomidine During Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MD ∕ 15.08.78
Record Dates: First submitted 2017-08-26; First posted 2017-08-29 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Radical Cystectomy
MeSH Terms: interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Experimental): Patients received intravenous infusion of dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- Fentanyl (Active Comparator): Patients received intravenous infusion of fentanyl
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive Loading dose of dexmedetomidine (0.8μg/kg) over 20 minutes, followed by intravenous infusion (0.4μg/kg/h) during intra-operative period till end of procedure.
  Arms: Dexmedetomidine
Drug: Fentanyl — Patients will receive Loading dose of fentanyl (1μg/kg), followed by intravenous infusion (1μg/kg/h) during intra-operative period till end of procedure.
  Arms: Fentanyl

SUMMARY:
Acute kidney injury and chronic kidney disease usually associated with radical cystectomy operation which is the treatment of choice for invasive urinary bladders tumor. Peri-operative acute kidney injury (AKI) is common but poorly recognized and managed which is associated with increase surgical morbidity and mortality and hospital cost .Prospective human studies establishing a renal protective effect of dexmedetomidine are still questionable.

DETAILED DESCRIPTION:
The aim of this study is to test the hypothesis that intra-operative intravenous dexmedetomidine infusion could improve early renal function after open radical cystectomy.

This randomized comparative study will be carried out on 100 patients of either sex, ASA I and II with baseline serum creatinine below 1.4 mg/dl who will be submitted for radical cystectomy. The patients will be randomly allocated into two groups according to the drug infused intra-operatively; dexmedetomidine group and fentanyl group. Dexmedetomidine group: will receive loading dose (0.8μg/kg) over 20 minutes, followed by intravenous infusion (0.4μg/kg/h) and fentanyl group: will receive loading dose (1μg/kg), followed by intravenous infusion (1μg/kg/h) during intra-operative period till end of procedure. Assessment of renal function through evaluation of pre-operative estimated glomerular filtration rate (eGFR) using Modification of Diet in Renal Disease (MDRD) formula based on baseline serum creatinine, serum cystatin C level at 24 hours post-operative, daily post-operative serum creatinine for one week post-operative and post-operative eGFR using MDRD formula.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I or II.
* Patients scheduled for elective radical cystectomy.

Exclusion Criteria:

* Serum creatinine level equal or greater than 1.4 mg/dl.
* Allergy to alpha-2 adrenergic agonist
* Allergy to any anesthetic drugs
* Uncontrolled hypertension.
* Uncontrolled diabetes.
* Heart block greater than first degree.
* History of alcohol abuse.
* History of drug abuse.
* Clinically significant neurologic disease.
* Clinically significant cardiovascular disease.
* Clinically significant respiratory disease.
* Clinically significant hepatic disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Serum cystatin C level | For 24 hours after surgery

SECONDARY OUTCOMES:
Serum creatinine | For 7 days after surgery
  Daily morning over the first post-operative week
Post-operative eGFR | For 7 days after surgery
  daily within the first week post-operative
Heart rate | For 8 hours after induction of general anesthesia
  recorded immediately after intubation, every 30 min during surgery and immediately after closure of the skin
Mean arterial blood pressure | For 8 hours after induction of general anesthesia
  recorded immediately after intubation, every 30 min during surgery and immediately after closure of the skin
Peripheral oxygen saturation (SpO2) | For 8 hours after induction of general anesthesia
  recorded immediately after intubation, every 30 min during surgery and immediately after closure of the skin
End-tidal carbon dioxide tension | For 8 hours after induction of general anesthesia
  recorded immediately after intubation, every 30 min during surgery and immediately after closure of the skin
Total volume of crystalloid solutions used | For 8 hours after induction of general anesthesia
  recorded immediately after intubation, every 30 min during surgery and immediately after closure of the skin
Total volume of colloid solutions used | For 8 hours after induction of general anesthesia
  recorded immediately after intubation, every 30 min during surgery and immediately after closure of the skin
Total volume of packed red blood cells transfused | For 8 hours after induction of general anesthesia
  recorded immediately after intubation, every 30 min during surgery and immediately after closure of the skin
Intraoperative occurrence of hypotension | For 8 hours after induction of general anesthesia
  recorded immediately after intubation, every 30 min during surgery and immediately after closure of the skin
Intraoperative occurrence of bradycardia | For 8 hours after induction of general anesthesia
  recorded immediately after intubation, every 30 min during surgery and immediately after closure of the skin

CONTACTS AND LOCATIONS:
Overall Officials: Golinar E Hammouda, MD, Study Chair — Department of Anaesthesia, Surgical Intensive Care and Pain Medicine, College of Medicine, Mansoura University, Mansoura, Egypt
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided